CLINICAL TRIAL: NCT02940665
Title: Higher Protein Intakes Are Associated With Reduced Length of Stay: A Comparison Between ERAS and Conventional Care After Elective Colorectal Surgery
Brief Title: A Comparison of Protein Intake Between ERAS and Conventional Care After Elective Colorectal Surgery
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: Canadian Foundation for Dietetic Research (CFDR) (Other)
Responsible Party: Principal Investigator, Dr. Tanis Fenton, Associate Professor, University of Calgary
Other Study IDs: 13-1337
Record Dates: First submitted 2016-10-14; First posted 2016-10-21 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Disorders; Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Enhanced Recovery After Surgery (ERAS): ERAS group followed the ERAS protocol. The protocol was implemented 13 months prior to the start of data collection.
  Interventions: Other: ERAS
- Conventional: Conventional group received conventional care.

INTERVENTIONS:
Other: ERAS — Patients in the ERAS group received the ERAS protocol
  Groups: Enhanced Recovery After Surgery (ERAS)

SUMMARY:
The primary objective of this prospective cohort study is to compare protein intake and adequacy between patients receiving Enhanced Recovery After Surgery (ERAS) protocols with patients receiving conventional care. The study will also compare energy intakes, gut function, and clinical outcomes between groups. The ability of nutritional parameters, including preoperative malnutrition risk and postoperative protein intake, to predict length of hospital stay will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* adult patients ≥18 years of age
* elective colorectal resection

Exclusion Criteria:

* co-morbidities that could have interfered with oral intake (e.g., dysphagia)
* concurrent enteral or parenteral nutrition prior to surgery were excluded since food intakes could be influenced by these conditions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Colorectal surgery
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Total protein intake (grams) as assessed by food records. | Average in first three postoperative days
  Protein intake from food records on postoperative days 1, 2 and 3 will be recorded. Patients will record the amount of food, fluid, and oral nutrition supplements consumed using quartiles (none, ¼, ½, ¾, all) on a food record. Research staff will verify the self-reported food records with the patients after each meal. Total protein intake in grams will be determined by comparing actual food intake (obtained from the food records) to the food composition records of our institution.

SECONDARY OUTCOMES:
Length of hospital stay (number of days) | Number of days spent in hospital during admission for surgery up to 6 months
  Total length of hospital stay will be recorded in days beginning at admission for surgery until discharge.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yeung SE, Hilkewich L, Gillis C, Heine JA, Fenton TR. Protein intakes are associated with reduced length of stay: a comparison between Enhanced Recovery After Surgery (ERAS) and conventional care after elective colorectal surgery. Am J Clin Nutr. 2017 Jul;106(1):44-51. doi: 10.3945/ajcn.116.148619. Epub 2017 May 3. PMID 28468890